CLINICAL TRIAL: NCT00414193
Title: Piperacillin/Tazobactam for Bacteremia With Organisms Producing Chromosomally-Encoded AmpC Beta-Lactamase
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Japan Health Sciences Foundation (Unknown)
Responsible Party: Principal Investigator, Yohei Doi, MD, University of Pittsburgh
Other Study IDs: IRB#0611104
Record Dates: First submitted 2006-12-19; First posted 2006-12-21 (Estimated); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Bacteremia; AmpC Beta-lactamase
Keywords: AmpC beta-lactamase; Bacteremia; Piperacillin; Tazobactam
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — No genetic testing will be performed on any of the samples being obtained. The biologic samples will be under the control of the principal investigator of this research project. To protect confidentiality, all personal identifiers (i.e., name, social security number, and birth date) will be removed (de-identified) and replaced with a specific code number. The information linking these code numbers to the corresponding subjects' identities will be kept in a separate, secure location. The investigators on this study will keep the samples indefinitely. If a subject withdraws and provides the request in writing, samples collected and not already processed will be destroyed. All samples will be kept in the investigator's laboratory located in Scaife Hall, Room 812, 3550 Terrace Street.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Nosocomial bloodstream infections are important causes of morbidity and mortality caused by AmpC beta-lactamase-producing Enterobacteriaceae. The information collected will optimize the management of patients with nosocomial bloodstream infections.

DETAILED DESCRIPTION:
The following information will be collected: age, sex, occupation, hospital location at the time of positive culture (ER, medical ward, ICU etc), prior hospitalization, receipt of outpatient dialysis, home care or other regular medical care (eg, outpatient chemotherapy), presence of invasive devices, receipt of antibiotics, including their type and whether they were adequate for the resistance profile of the organism, prior positive microbiologic cultures, time and location of positive cultures, underlying diseases and severity of illness, presence of urinary or intravascular devices, recent immunomodulative therapies or radiation therapy, physical exam findings, laboratory and radiographical data, antimicrobial usage within 30 days of onset of the infection, microbiological data and resistance patterns, choice of antibiotics once organism identified, bacteriological outcomes, laboratory results, demographic information, medications, clinical outcome,gender, height, weight, ethnicity, and past medical history. We will collect information retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Clinical information is collected by chart review of "case" and "control" patients. A "case" patient is defined as follows:

  * One or more blood cultures are positive for E. cloacae, E. aerogenes, C. freundii, S. marcescens or M. morganii.
  * The patient received piperacillin/tazobactam as the initial empiric therapy.
  * The organism was susceptible to piperacillin/tazobactam.
* A "control" patient is defined as follows:

  * One or more blood cultures are positive for E. cloacae, E. aerogenes, C. freundii, S. marcescens or M. morganii.
  * The patient received a carbapenem or fluoroquinolone antimicrobial as the initial empiric therapy.
  * The organism was susceptible to the empiric regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: positive cultures
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2007-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
dead or alive | end of study
  health status

CONTACTS AND LOCATIONS:
Overall Officials: David L Paterson, MD, Principal Investigator — University of Pitttsburgh; Yohei Doi, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States